CLINICAL TRIAL: NCT03000205
Title: Effects of Hypertonic Dextrose Water Injection for Supraspinatus Tendinosis Patients: Analysis of Clinical and Sonographic Presentation
Brief Title: Effects of Hypertonic Dextrose Water Injection for Supraspinatus Tendinosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201605022
Record Dates: First submitted 2016-10-11; First posted 2016-12-21 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2022-10

CONDITIONS: Chronic Shoulder Pain
Keywords: Dextrose prolotherapy; patients
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypertonic dextrose water (Experimental): 20% hypertonic dextrose water injection for chronic shoulder spin
  Interventions: Device: hypertonic dextrose water
- Normal Saline (Placebo Comparator): normal saline and Lidocaine as placebo for sham group
  Interventions: Device: Normal saline and Lidocaine.

INTERVENTIONS:
Device: hypertonic dextrose water — 20% hypertonic dextrose water injection for chronic shoulder pain at Week0
  Other Names: Prolotherapy group
  Arms: hypertonic dextrose water
Device: Normal saline and Lidocaine. — Normal Saline injection for chronic shoulder pain at Week0 (Arms:Placebo Comparator: Placebo)
  Other Names: Control group
  Arms: Normal Saline

SUMMARY:
Using hypertonic dextrose water for chronic supraspinatus tendinosis and using ultrasound as assessment tool to evaluate the effect of intervention.

DETAILED DESCRIPTION:
Supraspinatus tendinosis is a degenerative process of tendon. It can be caused by external trauma episode and imbalanced of self-repair process. It can cause patients with shoulder pain when shoulder over head exercise and heavy lifting. It can also influence the sleep quality due to pain symptoms of shoulder. Usually these patients had limited response to medication and physical modality. Moreover, it can cause shoulder tear or rupture, which can disability with aging. Prolotherapy is an injection therapy for chronic painful musculoskeletal conditions. It involves the injection of small volumes of an irritant agent, most commonly a hyperosmolar dextrose solution, at multiple painful tendon and ligament insertions where they connect to bone, over several treatment sessions. The injection of an irritant solution initiates an inflammatory cascade at the site of injection, which causes fibroblast proliferation and subsequent collagen synthesis, resulting in a stronger tendon or ligament. Hyperosmolar dextrose appears to be the most commonly used agent today, with morrhuate sodium used slightly less often. There is promising recent evidence for prolotherapy, with hyperosmolar dextrose in treating painful tendinopathies. The aim of this study is to hypertonic injection in supraspinatus tendinosis patients about clinical and ultrasound image presentation. We conducted a double blinded randomized controlled trial for 60 participants with chronic shoulder pain for 3 months with supraspinatus tendonsis. In study group, one injection with 20% dextrose water was injection in supraspinatus tendon and control group received normal saline and Lidocaine. SPADI, VAS and ultrasound data were obtained before intervention and 2 weeks, 6 weeks and 12 weeks after injection after intervention. The ANOVA and independent t test are applied for analysis by SPSS 20.0 with P value less than 0.05 as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 20 years old with diagnosis of chronic supraspinatus tendinosis by ultrasound and clinical shoulder pain lasting for more than 3 months

Exclusion Criteria:

* History of shoulder fracture and operation, with frozen shoulder or full thickness rupture of rotator cuff, steroid, or hyaluronic acid, or platelet rich plasma (PRP) injection during the period of intervention and following up

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2020-07 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Shoulder Pain and Disability Index (change of SPADI) | Week0 Week2 Week6 Week12
  Shoulder Pain and Disability Index (SPADI), a self-administered assessment tool that was used to measure pain and disability related to shoulder disease. The SPADI consists of 5 pain and 8 disability items that are measured on a visual analog scale. Pain and disability subscales were calculated as the mean of the corresponding items on a 0-100 scale; the highest score indicated the most severe pain and disability. The total outcome score used for statistical analysis was calculated as the sum of the pain and disability subscales.

SECONDARY OUTCOMES:
Ultrasound | Week0 Week2 Week6 Week12
  The ultrasound evaluated the status of the biceps and supraspinatus patency was evaluated using both longitudinal and transverse views. The findings of the ultrasound examinations were classified as either normal or abnormal (tear or tendonitis). A tear was defined as a discontinuity in the normal homogeneous echogenicity of the tendon, whereas tendonitis was defined as a thickening or hypoechogenicity of the tendon in the absence of a border defect. The diagnostic criteria of biceps tenosynovitis was defined as tendon sheath fluid accumulation (abnormal hypoechoic or anechoic accumulation relative to subdermal fat; occasionally isoechoic or hyperechoic) in intra-articular material that is displaceable and compressible at ≥ 3 mm.
Shoulder ROM (Range of Motion) | Week0 Week2 Week6 Week12
  Pain-free passive range of motion (PROM) of the shoulder was designated as the range of motion attained at the most painful position and was measured using a digital goniometer in 6 directions flexion, extension, abduction, adduction, external rotation and internal rotation. Five directions of the shoulder joint were measured (flexion, abduction, adduction, internal rotation, and external rotation) while participants were lying in a supine position. Additionally, shoulder extension was measured in the side-lying position.
Pain (VAS, Visual Analogue Scale) | Week0 Week2 Week6 Week12
  Shoulder pain was assessed according to an 11-point numerical rating scale (NRS). This tool was simple to use and was highly correlated with the visual analog scale, verbal rating scale, and Faces Pain Scale-Revised. The NRS is considered a valid and reliable pain assessment tool. The pain intensity was graded from 0 (no pain) to 10 (the most intense level of pain). The participants reported their pain level at rest and during the movement of shoulder joint in all direction. The most painful movement score was used for further data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, New Taipei City, Zhonghe Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No